Title: Protocol For Sleep for Critically III Patients

Date: 08/02/2023

NCT: 5.882.443

INFORMED CONSENT FORM IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE UNITS

You are being invited to participate in the research titled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital Moinhos de Vento. By agreeing to participate in this study, you will be asked to complete a questionnaire about the sleep quality in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed.

Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your treatment.

Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality.

If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000.

After reading this form in its entirety, I, \_\_\_\_\_\_\_, declare that I have understood the objectives of the study "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which will be conducted by researcher Laura Drehmer. I also declare that I have received a copy of this Informed Consent Form, with another copy remaining with the researcher, and that I agree to participate voluntarily in this research.

| Participant's signature: | - |
|--------------------------|---|
| Researcher's signature: | |

INFORMED CONSENT FORM

IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE UNITS

You are being invited to participate in the research titled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital da Unimed Vale dos Sinos. By agreeing to participate in this study, you will be asked to complete a questionnaire about the sleep quality in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed.

Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your treatment.

Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality.

If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000.

After reading this form in its entirety, I, \_\_\_\_\_\_\_, declare that I have understood the objectives of the study "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which will be conducted by researcher Laura Drehmer. I also declare that I have received a copy of this Informed Consent Form, with another copy remaining with the researcher, and that I agree to participate voluntarily in this research.

| Participant's signature: |
|---------------------------------------------------|
| Researcher's signature: |
| NFORMED CONSENT FORM FOR HEALTHCARE PROFESSIONALS |

IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE **UNITS** You are being invited to participate in the research titled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital Moinhos de Vento. By agreeing to participate in this study, you will be asked to complete a questionnaire about your perception regarding the sleep quality in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed. Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your treatment. Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality. If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000. After reading this form in its entirety, I, \_\_\_\_\_\_, declare that I have understood the objectives of the study "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which will be conducted by researcher Laura Drehmer. I also declare that I have received a copy of this Informed Consent Form, with another copy remaining with the researcher, and that I agree to participate voluntarily in this research.

Participant's signature: \_\_\_\_\_

Researcher's signature: \_\_\_\_\_\_

IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE UNITS

You are being invited to participate in the research titled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital da Unimed Vale do Sinos. By agreeing to participate in this study, you will be asked to complete a questionnaire about your perception regarding the sleep quality in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed.

Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your treatment.

Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality.

If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000.

| After reading this form in its entirety, I,, de | eclare |
|---|---|
| that I have understood the objectives of the study "MULTIDISCIPLII | NARY |
| PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which | h will |
| be conducted by researcher Laura Drehmer. I also declare that I have recei | ved a |
| copy of this Informed Consent Form, with another copy remaining wit | h the |
| researcher, and that I agree to participate voluntarily in this research. | |

| Participant's signature: <sub>-</sub> |
|---------------------------------------|
| Researcher's signature: |

## INFORMED CONSENT FORM FOR PATIENTS' FAMILY MEMBERS

IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE UNITS

You are being invited to participate in the research titled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital Moinhos de Vento. By agreeing to participate in this study, you will be asked to complete a questionnaire about your perception regarding the sleep quality of your family member in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed.

Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your family member's treatment.

Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality.

If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000.

| After reading this form in its entirety, I, | , declare |
|---|---|
| that I have understood the objectives of the study "MULTIDISCI | PLINARY |
| PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," w | vhich will |
| be conducted by researcher Laura Drehmer. I also declare that I have re | eceived a |
| copy of this Informed Consent Form, with another copy remaining | with the |
| researcher, and that I agree to participate voluntarily in this research. | |

| researcher, and that I agree to participate voluntarily in this research. |
|---------------------------------------------------------------------------|
| Participant's signature: |
| Researcher's signature: |

## INFORMED CONSENT FORM FOR PATIENTS' FAMILIES

IMPLEMENTATION PROJECT OF THE SLEEP PROTOCOL IN INTENSIVE CARE UNITS

You are being invited to participate in the research entitled "MULTIDISCIPLINARY PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," which aims to evaluate the effectiveness of an institutional protocol of actions to improve the sleep quality of patients admitted to the Intensive Care Units (ICU) at Hospital da Unimed Vale dos Sinos. By agreeing to participate in this study, you will be asked to complete a questionnaire about your perception regarding the sleep quality of your family member in the ICU, which aims to assess the implementation of a sleep protocol for patients. The benefits of this study may be perceived in the near future when, based on the analysis of your responses, action plans for continuous improvement of sleep quality in the ICU can be developed.

Participation in this study is entirely voluntary and will not incur any additional costs. Additionally, accepting this invitation will not entitle you to any remuneration. Even after agreeing to participate, you have the right and freedom to withdraw your consent at any stage of the research, regardless of the reason, without any prejudice to you or your family member's treatment.

Your participation in the study will be entirely voluntary and anonymous. You will not be identified in any way. The risks related to your participation include the time spent responding to the questionnaire and the risk of a breach of confidentiality.

If you have any doubts, you can clarify them by contacting researcher Laura Drehmer at phone (51) 9998867-22, Dr. Felipe Dexheimer at phone (51) 991195508, or the Ethics and Research Committee of Hospital Moinhos de Vento, by phone (51) 33143537, located at Rua Ramiro Barcelos, 910, 4th floor – Building A, Bairro Floresta, Porto Alegre, RS, Brazil, ZIP Code 90035-000.

| After reading this form in its entirety, I, | , declare |
|---|---|
| that I have understood the objectives of the study "MULTIDISCI | PLINARY |
| PROTOCOL FOR IMPROVING SLEEP QUALITY IN CRITICAL PATIENTS," w | hich will |
| be conducted by researcher Laura Drehmer. I also declare that I have re | eceived a |
| copy of this Informed Consent Form, with another copy remaining | with the |
| researcher, and that I agree to participate voluntarily in this research. | |

| Participant's signature: | <br>_ |
|--------------------------|-------|
| Researcher's signature: | |